CLINICAL TRIAL: NCT06083922
Title: A Phase II Study of CyBorD (Cyclophosphamide, Bortezomib, Dexamethasone) Plus Daratumumab for Patients With Monoclonal Gammopathy of Renal Significance (MGRS)
Brief Title: A Study of CyBorD (Cyclophosphamide, Bortezomib, Dexamethasone) Plus Daratumumab in People With Monoclonal Gammopathy of Renal Significance (MGRS)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Janssen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 22-424
Record Dates: First submitted 2023-10-06; First posted 2023-10-16 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Multiple Myeloma; Monoclonal Gammopathy of Renal Significance
Keywords: Cyclophosphamide; Bortezomib; Dexamethasone; Daratumumab; 22-424
MeSH Terms: conditions — Multiple Myeloma | interventions — Cyclophosphamide; Bortezomib; Dexamethasone; daratumumab

STUDY DESIGN:
Intervention Model Description: This trial will include a safety run-in-stage that will enroll patients from either cohort, which purpose is to test the safety of the combination. The run-in-stage will be followed by:
  A Simon-two-stage phase II study that will enroll patients with cast nephropathy (cohort A), A pilot study that will enroll patients with all other MGRS excluding AL amyloidosis (cohort B).
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A will include patients with cast nephropathy (Experimental): Planned 8 cycles of CyBorD-Dara SC, treatment will be left to the discretion of the treating physician. It is recommended that patients eligible for ASCT undergo ASCT after 8 cycles of induction and that patient ineligible for ASCT, continue maintenance Bortezomib/Dexamethasone administered every other week with daratumumab SC administered every 4 weeks, for a period of 2 years from start of treatment.
  Interventions: Drug: Cyclophosphamide; Drug: Bortezomib; Drug: Dexamethasone; Drug: Daratumumab
- Arm B will include all other MGRS associated diseases with the exclusion of AL amyloidosis (Experimental): Planned 8 cycles of CyBorD-Dara SC, treatment will be left to the discretion of the treating physician. It is recommended that patients eligible for ASCT undergo ASCT after 8 cycles of induction and that patient ineligible for ASCT, continue maintenance Bortezomib/Dexamethasone administered every other week with daratumumab SC administered every 4 weeks, for a period of 2 years from start of treatment.
  Interventions: Drug: Cyclophosphamide; Drug: Bortezomib; Drug: Dexamethasone; Drug: Daratumumab

INTERVENTIONS:
Drug: Cyclophosphamide — Days 1, 8 and 15, Cycles 1-8
Drug: Bortezomib — Days 1,8,15, Cycles 1-8, Days 1,15 Cycles 9+
Drug: Dexamethasone — Days 1,2,8, 9,15,16, 22, 23, Cycles 1-8
Drug: Daratumumab — Days 1,8,15,22, Cycles 1-2, Days 1,15 Cycles 3-6, Day 1 Cycles 7+

SUMMARY:
The purpose of this study is to find out whether cyclophosphamide, bortezomib, dexamethasone (CyBorD) with daratumumab SC is a safe treatment combination for MGRS-associated kidney disease including cast nephropathy associated with multiple myeloma. In addition, the researchers will find out whether the study drug combination is an effective treatment for these conditions.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for cast nephropathy associated with MM:

* Subjects must have a confirmed diagnosis of NDMM as per standard IMWG criteria
* Subjects must have measurable disease, defined as meeting at least 1 of the following criteria ≤ 14 days prior to registration:

  * A monoclonal Immunoglobulin (M-protein) concentration on serum protein electrophoresis (SPEP) of ≥ 0.5 g/dL.
  * Measurable urinary light chain secretion by quantitative analysis using urine protein electrophoresis (UPEP) of ≥ 200 mg/24 hours.
  * Involved serum free light chain (FLC) level ≥ 10 mg/dL, provided the serum FLC ratio is abnormal.
* eGFR must be <40 ml/min/1.73m2
* Subjects must have histologically confirmed diagnosis of monoclonal gammopathy associated CN by kidney biopsy OR If a kidney biopsy is not available, a percentage of urine albumin excretion (%UAE) < 25 % AND FLC > 50 mg/dL

Inclusion criteria for other MGRS associated renal diseases

* Histologically confirmed diagnosis of MGRS-associated renal disease by kidney biopsy
* Presence of monoclonal gammopathy by serum protein electrophoresis, Immunofixation, or Free Light Chain Assay
* Evidence of plasma cell dyscrasia by bone marrow biopsy confirming clonal plasma cell population
* eGFR <40 ml/min/1.73m2 or 24h urine total protein > 1gm

Inclusion criteria for both cast nephropathy associated with MM and other MGRS associated renal diseases

* Subjects must be ≥ 18 years of age at time of registration.
* Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 ≤ 14 days prior to registration.
* No evidence of unequivocal recent nephrotoxic exposure (NSAIDs, radiocontrast…)
* No evidence of obstructive nephropathy by ultrasound
* Subjects must have adequate hematology laboratory values within 14 days prior to registration defined by the following:

  * Neutrophils ≥ 1.0 × 10^9 /L (Patients cannot have received G-CSF or GM-CSF within 1 week of screening or pegfilgrastim within 2 weeks of screening to meet eligibility).
  * Platelets ≥ 100 × 10^9 /L for run-in and 75 × 10^9 /L for phase II (Note: Platelet support is not permitted to help participants meet eligibility criteria).
  * hemoglobin ≥ 7.5 g/dL without prior red blood cells [RBC] transfusion within 7 days before the laboratory test; recombinant human erythropoietin use is permitted.
* Subjects must have adequate hepatic function laboratory values ≤ 14 days prior to registration:

  * Aspartate aminotransferase (AST), alkaline phosphatase (AP) or alanine aminotransferase (ALT) ≤ 3 × the upper limit of normal (ULN)
  * Total bilirubin ≤ 1.5 x ULN except for patients with a history of elevated total bilirubin, such as in Gilbert's.
  * Hepatic Child-Pugh score at worse A (patients are eligible for the phase 2 part but not for the Run-in-Period of the trial).
* Female patients will have to satisfy the following criteria:

  * Be postmenopausal for at least 1 year Prior to registration visit, OR
  * Be surgically sterile, OR
  * If of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception). If patient is female and of childbearing potential, she must have a negative serum beta human chorionic gonadotropin (β-HCG) test < 14 days prior to registration and consent to ongoing pregnancy testing during the course of the study.
* Male patients, even if surgically sterilized (i.e., status post-vasectomy), must agree to one of the following

  * Practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR
  * Practice true abstinence when this is in line with the preferred and usual lifestyle of he subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable methods of contraception).
* Subjects must have the willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, study procedures, and research procedures.

Exclusion Criteria:

* MGRS associated with diseases other than plasma cell dyscrasia (e.g. CLL, B-cell neoplasm, Waldenstrom's macroglobulinemia…)
* Plasma cell leukemia, AL amyloidosis, or POEMS syndrome.
* Treatment with prior drugs aimed at the plasma cell dyscrasia.
* Treatment with prior or concurrent investigational agents aimed at the plasma cell dyscrasia.
* Female patients who are lactating or have a positive serum pregnancy test during the screening period.
* Major surgery ≤ 14 days before registration.
* Focal radiation therapy within 14 days prior to registration with the exception of palliative- radiotherapy for symptomatic management but not on measurable extramedullary plasmacytoma.
* Disease-related central nervous system involvement.
* The subject has uncontrolled significant intercurrent illness including, but not limited to, ongoing or active infection.
* Clinically significant cardiac disease, including:

  * Myocardial infarction within 6 months before randomization, or unstable or uncontrolled disease/condition related to or affection cardiac function (e.g., unstable angina, congestive heart failure, New York Heart Association Class III-IV)
  * Uncontrolled cardiac arrhythmia
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
* Concurrent malignancy except for treated non-melanoma skin cancer, cervical carcinoma in situ and low-risk prostate CA being monitored without treatment.
* Grade 2 or higher peripheral neuropathy on clinical examination during the screening period.
* Chemotherapy ≤ 14 days of registration.
* Exposure to an investigational drug (including investigational vaccine) or invasive investigational medical device for any indication within 4 weeks or 5 pharmacokinetic halflives, whichever is longer.
* Patients with known chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) <50% of predicted normal; moderate or severe persistent asthma within the past 2 years. Note that FEV1 testing is required for participants suspected of having COPD and participants must be excluded if FEV1 is <50% of predicted normal
* Moderate or severe persistent asthma within the past 2 years, or uncontrolled asthma of any classification. Note that participants who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed to participate.
* Patients who have a contraindication to the use of any form of anticoagulation or antiplatelet agents.
* The use of strong CYP3A4 and CYP1A2 inducers or inhibitors will not be allowed while patients are treated on this study.
* Patients with Hepatic Child-Pugh score B and C. Note that patients with Hepatic Child-Pugh score A are excluded from the Run-in-Period of the trial
* Patient is:

  * Known history of human immunodeficiency virus (HIV) and those who are seropositive for HIV.
  * Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Subjects with resolved infection (ie, subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR.
  * Seropositive for hepatitis C (except in the setting of a sustained virologic response [SVR], defined as aviremia at least 12 weeks after completion of antiviral therapy).
  * Vaccination with live attenuated vaccines within 4 weeks of first study agent administration.
  * Plasmapheresis within 28 days before randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Run-in Phase- Dose-limiting toxicity (DLT) rates | 2 years
  Any participant in the run-in-phase who received at least ≥ 75% of the planned doses of the combination regimen in cycle one will be evaluated for DLTs using NCI-CTCAE.
Phase II (Cohort A) best renal response | 2 years
  For patients with a decreased eGFR <50mL/min/1.73 m2 with or without significant proteinuria (UTP>0.5 gm/24h) at presentation, Assessment of renal response will be based on both the IMWG criteria for patient with decreased eGFR and the amyloid criteria for patients with proteinuria.
Pilot study (Cohort B) best renal response | 2 years
  For patients with a decreased eGFR <50mL/min/1.73 m2 with or without significant proteinuria (UTP>0.5 gm/24h) at presentation, renal response will be assessed using IMWG renal response criteria

CONTACTS AND LOCATIONS:
Overall Officials: Hani Hassoun, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (11):
- United States (11):
  - Tufts Medical Center (Data Collection Only), Boston, Massachusetts
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Weill Cornell Medical Center (Data Collection Only), New York, New York
  - Mount Sinai Hospital (Data Collection Only), New York, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York
  - University of North Carolina (Data Collection Only), Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm